CLINICAL TRIAL: NCT05901844
Title: Evaluate the Effectiveness and Safety of the Raman IVD Analyzer for Intraoperative Glioma Diagnosis, Using Samples From Brain Resection Tissue (Prospective, Multicenter, Blind Evaluation, Single Group Target Value Method)
Brief Title: Evaluate the Accuracy of Raman IVD Analyzer in the Diagnosis of Gliomas During Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: West China Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Capital Medical University (Other); Jiangsu Raman Medical Equipment Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LRR202301
Record Dates: First submitted 2023-05-24; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Glioma
Keywords: glioma; Raman; intraoperative; surgery
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Intervention Model Description: The same sample was diagnosed using Raman spectroscopy and paraffin pathology, respectively. Calculate the sensitivity and specificity of a Raman analyzer using paraffin pathological results as the gold standard.
Masking Description: Blind assessment: Researchers using Raman analyzer during surgery are not aware of the subjects' preoperative diagnostic results, while researchers conducting paraffin pathology examinations after surgery are not aware of the subjects' preoperative diagnostic results and the diagnostic results of Raman analyzer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perform two different tests on the same sample (Other): The same sample is diagnosed using a Raman analyzer firstly and then diagnosed by paraffin pathology.
  Interventions: Diagnostic Test: Paraffin pathological diagnosis

INTERVENTIONS:
Diagnostic Test: Paraffin pathological diagnosis — Perform two diagnostic methods on the same sample
  Other Names: Raman analyzer diagnosis

SUMMARY:
Compare the data obtained from the Raman analyzer and paraffin pathology examination on the same external brain tissue sample. Evaluate the effectiveness and safety of the Raman analyzer for intraoperative diagnosis gliomas of brain resection tissue samples, using paraffin pathological examination results as clinical reference standards.

DETAILED DESCRIPTION:
Based on statistical calculations,108 positive samples and 148 negative samples will be included in the trial in all trial centers. Compare the results between the Raman analyzer and the paraffin pathological. And calculate the sensitivity, the specificity, and other indicators of Raman analyzer.

During surgery, core or marginal tissue samples were taken from subjects. The test samples size:0.2cm<length diameter ≤ 2cm. The sample testing result is based on the Raman test points. Then take the same tissue sample for paraffin pathological diagnosis.

Statistical description of all data, including baseline data, all efficacy indicators, and all safety data. The measurement data give the mean, standard deviation, minimum, maximum, median,25 quantile and 75 quantile; Provide frequency and composition ratio for counting data. The baseline data was analyzed using the Full Analysis Set (FAS); The effectiveness analysis adopts FAS and PPS; The security analysis uses the Security Dataset (SS).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, regardless of gender;
* Patients who plan to undergo brain lesion tissue resection surgery or have preoperative clinical diagnosis of gliomas and plan to undergo biopsy;
* Patients with clinical diagnosis of initial solitary gliomas, or initial solitary intracranial masses or initial non occupying lesions that do not exclude gliomas (such as intracranial metastatic lesions, intracranial infectious lesions, intracranial demyelinating lesions, central nervous system lymphoma, etc.), who have not received radiotherapy or chemotherapy in the past based on their medical history;
* The patient or their guardian can understand the research purpose, demonstrate sufficient compliance with the trial protocol, and sign an informed consent form;
* It is possible to obtain tissue samples with a length diameter greater than 0.2cm. Patients diagnosed with initial solitary glioma should take core or marginal tissue, while patients diagnosed with initial single intracranial mass or initial non mass lesions but maybe with gliomas should be taken core tissue.

Exclusion Criteria:

* Investigator judge that it is not suitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the Raman analyzer in detecting gliomar | Through study completion, an average of 1 year
  Among the samples determined by paraffin pathology as gliomas, the percentage of samples detected by Raman analyzer as gliomas.
Specificity of the Raman analyzer in detecting gliomar | Through study completion, an average of 1 year
  Among the samples determined by paraffin pathology as non gliomas, the percentage of samples detected by the Raman analyzer as non gliomas.

SECONDARY OUTCOMES:
Using the paraffin test results as a reference, calculate the accuracy of the Raman analyzer in detecting gliomar | Through study completion, an average of 1 year
  The proportion of tissue samples with consistent results between Raman analyzer detection and paraffin pathological diagnosis.
Positive predictive value of the Raman analyzer in detecting gliomar | Through study completion, an average of 1 year
  The percentage of samples diagnosed with glioma by paraffin pathology in the samples detected as glioma by Raman analyzer
Negative predictive value of Raman analyzer in detecting gliomar | Through study completion, an average of 1 year
  The percentage of samples diagnosed with non glioma by paraffin pathology in the samples detected as non glioma by Raman analyzer
Kappa coefficient | Through study completion, an average of 1 year
  Kappa coefficient≥0.75 indicates high consistency; 0.75>Kappa coefficient≥0.4, considered consistent; If the Kappa coefficient is less than 0.4, it is considered inconsistent.
The Raman analyzer usability evaluation | Through study completion, an average of 1 year
  Use Evaluation Form
Time consumption for the Raman analyzer in detecting gliomar | Through study completion, an average of 1 year
  Time required from emitting laser to completing single point detection

OTHER OUTCOMES:
The defect occurrence rate of the Raman analyzer | Through study completion, an average of 1 year
  The proportion of subjects with defects in the Raman analyzer during normal use to the total number of subjects using the Raman analyzer
Adverse Event Incidence Rate | During the surgery
  Number of subjects with AE/total number of subjects ×100%
Serious Adverse Event Incidence Rate | During the surgery
  Number of subjects with SAE/total number of subjects ×100%
Operator adverse events | Through study completion, an average of 1 year
  Possible damage to device operators during the use and maintenance of the Raman analyzers

CONTACTS AND LOCATIONS:
Overall Officials: Tao Jiang, MD and PhD, Principal Investigator — Beijing Tiantan Hospital; Qing Mao, Principal Investigator — West China Hospital; Dongming Yan, Principal Investigator — The First Affiliated Hospital of Zhengzhou University; Shouwei Li, Principal Investigator — Capital Medical University